CLINICAL TRIAL: NCT05316714
Title: Novel Nanofat Regenerative Surgical Technique for Peyronies' Disease Treatment With Penile Lenght Conservation and Non-incisional Albuginea Preservation
Brief Title: Novel Nanofat Regenerative Surgical Technique for Peyronies' Disease Treatment
Acronym: IPPNANOFAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Antonio Luigi Pastore, Associate Professor, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPP_2022_NanoFAT
Record Dates: First submitted 2022-03-20; First posted 2022-04-07 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Peyronie Disease
MeSH Terms: conditions — Penile Induration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IPP Nanofat Grafting (Experimental): Nanofat surgical grafting in albuginea penile tunica
  Interventions: Procedure: Nanofat grafing

INTERVENTIONS:
Procedure: Nanofat grafing — NANOFAT REGENERATIVE SURGICAL GRAFTING IN PRNILE ALBUGIANEA OF PATIENTS AFFECTED BY PEYRONIES' DISEASE

SUMMARY:
Peyronies' disease (PD) is an acquired connective tissue disorder characterized with the growth of fibrous and/or calcified plaques in the tunica albuginea of the penis.

The pathogenesis is still unclear, but the most accepted hypothesis is that in genetically prone individuals, trauma or repetitive microtraumas to the erect penis causes inflammation, and consequent growth of fibrous tissue due to degradation of the elastic fibers and fibrin deposition.

The fibrous plaques in the tunica albuginea of the penis causes typical signs and symptoms: penile abnormal curvature, penile pain, erectile dysfunction, indentation, loss of girth, shortening of the penis, with significant distress experience and psychological bother.

A lot of treatement have been proposed to date but with unsatisfactory results and the surgery results the definitive treatement but with possible risks.

Autologous fat grafting was first described by Neuber in 1893 and since then it has developed over the next century. The initial goal of fat grafting was to treat volume losses created by disease or trauma. Further studies done by Zuk et al. in 2001 showed that lipoaspirate contains multipotent adipose stem cells (ADSCs) like in the bone marrow, thereby expanding opportunities in multiple fields. ADSCs have emerged as a key element of regenerative medicine surgery due to their ability to differentiate into a variety of different cell lineages. Moreover, their capacity of paracrine secretion of a broad selection of cytokines, chemokines, and growth factors make them highly clinically attractive. More specific, of particular interest are the anti-apoptotic, anti-inflammatory, proangiogenic, immunomodulatory, and anti-scarring effects that have been demonstrated for ADSCs, which effects on wound healing, soft-tissue restoration and scar remodelling.

Nanofat firstly introduced by Tonnard in 2013, is an ultra-purified adipose tissue-derived product that is devoid of mature adipocytes but rich in ADSCs and with regenerative properties.

The aim of the study is to investigate the use of nanofat grafting in the treatement of PD.

DETAILED DESCRIPTION:
The etiology of PD remains uncertain, but is well accepted that there is a chronic inflammation of tunica albuginea and this reflect perturbations in normal wound healing and aberrant deposition of extracellular matrix components in the soft tissue of the penis.

There appears to be significant pathophysiologic and genetic overlap of PD with other superficial fibrosing disorders such as Dupuytren disease (palmar fibromatosis) and Ledderhose disease (plantar fibromatosis) but not with more diffuse conditions such as systemic sclerosis. Since PD was discovered, a lot of treatment were proposed. In the acute stage of PD treatments aim to alleviate penile pain and minimise disease progression and treatement attempts to mitigate inflammation: oral, intralesional injection, topical treatement were used but with few non significant results.

In the chronic phase, surgical treatments aims to correct the curvature but with not a few negative implications include penile shortening, erectile dysfunction, glans hypoaesthesia, residual or recurrent curvature and palpable or uncomfortable suture knots below the skin.

Recent findings on scar biology explain some factors that influence pro-fibrotic pathways. Preventions and treatment strategies mainly focus on reducing inflammation and hypoxia. Emerging therapies shows that Mesenchymal stem cells (MSCs) have immunomodulatory and antifibrotic effects by secreting paracrine growth factors.

Zuk et al. in 2001 and 2002 showed that lipoaspirate contains multipotent adipose stem cells (ADSCs) population comparable to that isolated from the bone marrow. Because of its availability and accessibility, white adipose tissue is considered a "stem cell depot." Nanofat grafting technique firstly reported by Tonnard is an ultra-purified adipose tissue-derived product that is devoid of mature adipocytes but contains rich in ADSCs, microvascular fragments, growth factors [vascular endothelial growth factor (VEGF), platelet-derived growth factor (PDGF), hepatocyte growth factor (HGF), transforming growth factor-beta (TGF-β), basic fibroblast growth factor (bFGF), insulin-like growth factor 1 (IGF-1), and granulocyte-macrophage colony-stimulating factor (GM-CSF)], biological peptides [lipoxins, resolvins, protectins, neurotrophic factors, angiogenin, matrix metalloproteinase, leukemia inhibitory factor, and macrophage migration inhibitory factor], and cytokines . It is a liquefied, autologous injectable product with the property of biological integration with adjacent cells and tissues due to its homogenous consistency. At the site of injury, these stromal cells initiate a site-specific reparative response comprised of remodeling of extracellular matrix, enhanced and sustained angiogenesis, immune system modulation, and cellular turnover. These properties of stromal cells provide a platform for the usage of cellular therapy in various diseases. Peyronie's "plaque" is a scarred tissue, results from abnormal extracellular matrix production through upregulation of myofibroblast activity and tissue inhibitors of matrix metalloproteinases, among other mechanisms. The aim of the study is to investigate the possible therapeutic role of nanofat grafting in the treatement of PD.

ELIGIBILITY:
Inclusion Criteria:

* Presence of albuginea penile plaque due to Peyronies' disease associated with penile curvature and pain. Normal erectile function. Sexual activity.

Exclusion Criteria:

* Erectile dysfunction, no sexual activity.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
Degree of curvature | Change from Baseline Penile curvature at 6 months
  Penile curvature assessment with in-office goniometric angle measurement of a pharmacologically induced erection
PAIN assessment | Change from Baseline PAIN (VAS SCORE) at 6 months
  Pain wil be assessed by VAT scale

CONTACTS AND LOCATIONS:
Locations (1):
- Antonio Luigi Pastore, Latina, Italy

IPD SHARING:
Plan to Share IPD: No
Outcomes

REFERENCES:
- [Result] Tonnard P, Verpaele A, Peeters G, Hamdi M, Cornelissen M, Declercq H. Nanofat grafting: basic research and clinical applications. Plast Reconstr Surg. 2013 Oct;132(4):1017-1026. doi: 10.1097/PRS.0b013e31829fe1b0. PMID 23783059
- [Result] Osmonov D, Ragheb A, Ward S, Blecher G, Falcone M, Soave A, Dahlem R, van Renterghem K, Christopher N, Hatzichristodoulou G, Preto M, Garaffa G, Albersen M, Bettocchi C, Corona G, Reisman Y. ESSM Position Statement on Surgical Treatment of Peyronie's Disease. Sex Med. 2022 Feb;10(1):100459. doi: 10.1016/j.esxm.2021.100459. Epub 2021 Nov 22. PMID 34823053